CLINICAL TRIAL: NCT02753361
Title: Ultrasound-Guided Regional Blockade for Lipoma Excision: a New Approach to an Old Technique
Brief Title: Ultra-sounded Guided Regional Blockade for Lipoma Excision
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Principal Investigator, Tarek F.Tammam, Tarek F.Tammam, M.D., Ph.D, Department of Anesthesia and Intensive Care, Faculty of Medicine, Suez Canal University Hospital, Egypt, Suez Canal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TTammam; Suez Canal University (Registry Identifier: Ghada A. Kamhawy)
Record Dates: First submitted 2016-04-24; First posted 2016-04-27 (Estimated); Last update posted 2017-10-19 (Actual); Status verified 2017-10

CONDITIONS: Lipomas
Keywords: Ultrasound; regional blockade; lipoma
MeSH Terms: conditions — Lipoma

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Traditional (No Intervention): This will utilize the traditional method of performance of regional block
- US-guided (Experimental): In this arm, regional block will be performed under the ultrasound guidance
  Interventions: Procedure: Ultrasound guidance

INTERVENTIONS:
Procedure: Ultrasound guidance — In the second arm, ultrasound will be used to guide the regional block
  Arms: US-guided

SUMMARY:
There is limited information on using the ultrasonography for block placement concerning lipoma excision. A new type of regional blockade, performed under ultrasound, can ensure proper block placement with accurate local anesthetics deposition. Investigators hypothesized that ultrasound guidance can reduce the number of needle passes to complete the block placement. Investigators will compare namely ultrasound guided regional blockade and traditional method regarding the number of needle passes to complete the block placement.

DETAILED DESCRIPTION:
50 patients between the ages of 18 and 60 years with American Society of Anesthesiologists (ASA) physical status I-III, scheduled for superficial subcutaneous lipoma (sized from 5 to 7 cm) excision will be enrolled in prospective comparative randomized clinical study.

Patients will be randomized into two groups: U (n = 25), in whom regional blockade was performed using US-guidance; and C (n = 25), in whom regional block was performed using the traditional method. Patients will be randomly assigned on a one-to-one ratio. Randomization will be performed by means of a computer generated random-numbers table. Group allocation will be concealed in sealed opaque envelopes that will not opened until patient consent had been obtained.

All patients will be pre-medicated with oral diazepam (7.5 mg) 30 min before the procedure, and IV fentanyl (50 ug) will be administered 5 minutes before placement of the block. Before the procedure, an IV access and standard monitoring of electrocardiogram (ECG), noninvasive blood pressure (NIBP), and peripheral oxygen saturation (SPO2) will be established.

Primary outcome includes the number of needle attempts (number of skin punctures and needle redirections) needed to complete the block placement. It will be documented by an investigator blinded to the aim of the study. Patient demographics, duration of surgery, patient's ASA physical status and other study outcomes will be documented by independent investigators who were not involved in the block placement procedure and were blinded to the group assignment.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 18 and 60 years
* American Society of Anesthesiologists (ASA) physical status I-III
* Superficial subcutaneous lipoma excision surgery (sized from 5 to 7 cm)
* Able to provide informed consent
* Consent to participates
* Single procedure

Exclusion Criteria:

* Unable to consent
* Do not consent to participate
* Patients with local infections in the skin over lipoma
* Patients with history of allergy to local anesthetics
* More than one procedure is being performed at the same setting

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2016-05; Primary Completion 2016-11-16 (Actual); Study Completion 2016-12-07 (Actual)

PRIMARY OUTCOMES:
The number of needle attempts needed to complete the block placement. New attempt will be defined as needle reinsertions through separate skin puncture. | 10 - 20 minutes

SECONDARY OUTCOMES:
The block success rate | 20 minutes
  The block success rate is assessed according to the adequacy of surgical anesthesia and is defined as complete loss of sensation to pinprick within 20 min of anesthetic administration and if no supplementation (sedative or analgesic) is required during surgery.Partial block is defined as inadequate sensory blockade after 20 min of anesthetic administration. The supplementation (additional LA infiltration or IV analgesic; fentanyl) is required to complete the proposed surgery. Failed block is considered if general anesthesia is required to complete the proposed surgery.
The incidence of adverse events | 8 hours postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Tarek F. Tammam, Prof., Study Director — Suez Canal university,Faculty of Medicine
Locations (1):
- Suez canal University hospital, Ismailia, Egypt

IPD SHARING:
Plan to Share IPD: Undecided